CLINICAL TRIAL: NCT04453917
Title: Dynamics of T Cell Expression of Immune Checkpoint Molecules in Progressive Multifocal Leukoencephalopathy
Acronym: ICIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/19/0506
Record Dates: First submitted 2020-06-03; First posted 2020-07-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: Progressive multifocal leukoencephalopathy; Pathophysiology; Immune checkpoint molecules; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal | interventions — Urination; Spinal Puncture

STUDY DESIGN:
Intervention Model Description: Patients with neurological symptoms (< 3 months) with brain MRI lesions suggestive of PML and positive PCR in cerebrospinal fluid for JCV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with active PML (Experimental): Patients with neurological symptoms (< 3 months) with brain MRI lesions suggestive of PML and positive PCR in cerebrospinal fluid for JCV
  Interventions: Biological: Collection of blood and urine; Biological: Spinal tap; Diagnostic Test: Brain MRI; Biological: Neurological evaluation

INTERVENTIONS:
Biological: Collection of blood and urine — Collection of blood (47 mL) and urine (5 mL) at PML diagnosis and 1, 3 and 6 months after, for analysis of immune checkpoint molecules expression, detection of antiviral immune responses and virological analyses.
Biological: Spinal tap — Spinal tap for monitoring of JC viral load at PML diagnosis and 1, 3 and 6 months after, and collection of CSF (2 mL) for virological analyses.
Diagnostic Test: Brain MRI — Brain MRI at at PML diagnosis and 3 and 6 months after
Biological: Neurological evaluation — Neurological evaluation at PML diagnosis and 1, 3 and 6 months after

SUMMARY:
Progressive multifocal leukoencephalopathy (PML) is a rare viral infection of the central nervous system (CNS) occurring in immunocompromised patients. Recovery of JC virus (JCV) specific T cell immune responses is the only available therapeutic option. JCV may use immune checkpoint inhibitory pathways to evade immune responses. The aim of this project is to determine whether T cell expression of immune checkpoint molecules is correlated to antiviral T cell responses, control of JCV replication and PML outcome. Immune checkpoint blockade by reversing T cell exhaustion may represent a therapeutic perspective for PML.

DETAILED DESCRIPTION:
PML is a devastating orphan disease of the CNS due to the reactivation of JCV in immunocompromised patients. Given the lack of drugs controlling JCV replication, initiation of antiretroviral therapy in HIV-infected patients or cessation of immunosuppressive therapies in others, and subsequent recovery of JCV-specific T cell immune responses remains to date the only available therapeutic option. Promoting antiviral immune responses may improve the control of viral replication and the outcome of this severe disease. Immune checkpoint molecules such as PD-1 are inhibitory receptors expressed on T cells that trigger inhibitory signaling pathways, limiting effector immune responses in cancer and chronic infections. Immune checkpoint inhibitory pathways implicated in evading immune responses may be at play in PML. Immune checkpoint blockade using monoclonal antibodies targeting PD-1, by reversing T cell exhaustion, has been suggested as a therapeutic perspective for PML. More insights in the dynamics of immune checkpoint molecules expressed by T cells in PML patients are needed to pave the way for a therapeutic study.

The aim here is to determine whether T cell expression of a broad range of immune checkpoint molecules, and its dynamics, correlates with the generation of antiviral of immune responses, the control of JCV replication and PML outcome.

To this end the investigators will recruit 15 PML patients from 4 teaching hospitals in the South West of France and assess at PML diagnosis and 1, 3 and 6 months after, the expression of immune checkpoint molecules on circulating T cells, ex vivo specific immune responses against a JCV peptide library, JC viral load in cerebrospinal fluid, blood and urine, and clinical and neuroradiological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old
* Informed consent
* Active virological PML : Recent neurological symptoms (< 3 months) with brain MRI lesions suggestive of PML and positive PCR in cerebrospinal fluid for JCV
* Affiliated or benefiting from public health insurance.

Exclusion Criteria:

* Non active PML
* Possible PML with negative JCV PCR
* Adults under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision
* Pregnant and/or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Immune checkpoint molecules | 1 month
  Expression level of a broad panel of immune checkpoint molecules by T cells at PML diagnosis bu flow cytometry
Immune checkpoint molecules | 3 months
  Expression level of a broad panel of immune checkpoint molecules by T cells at PML diagnosis bu flow cytometry
Immune checkpoint molecules | 6 months
  Expression level of a broad panel of immune checkpoint molecules by T cells at PML diagnosis bu flow cytometry
JC viral load | 1 month
  JC viral load in cerebrospinal fluid, blood and urine by ultra-sensitive PCR at PML diagnosis
JC viral load | 3 months
  JC viral load in cerebrospinal fluid, blood and urine by ultra-sensitive PCR at PML diagnosis
JC viral load | 6 months
  JC viral load in cerebrospinal fluid, blood and urine by ultra-sensitive PCR at PML diagnosis
Detection of immune responses against a JCV peptide library | 1 month
  Detection of specific immune responses against a JCV peptide library at PML diagnosis by flow cytometry
Detection of immune responses against a JCV peptide library | 3 months
  Detection of specific immune responses against a JCV peptide library at PML diagnosis by flow cytometry
Detection of immune responses against a JCV peptide library | 6 months
  Detection of specific immune responses against a JCV peptide library at PML diagnosis by flow cytometry

SECONDARY OUTCOMES:
Differential impact of immune checkpoint inhibition | 1 month, 3 months and 6 months
  Differential impact of immune checkpoint inhibition in vitro on detection of specific immune responses at PML diagnosis by flow cytometry
Clinical outcome with Performance status | 1 month, 3 months and 6 months
  Clinical outcome using validated scales such as Performance status at PML diagnosis
Clinical outcome with NIHSS | 1 month, 3 months and 6 months
  Clinical outcome using validated scales such as NIHSS (National Institute of Health Stroke Score) at PML diagnosis
Clinical outcome with Rankin | 1 month, 3 months and 6 months
  Clinical outcome using validated scales such as Rankin at PML diagnosis
Neuroradiological monitoring | 3 months and 6 months
  Neuroradiological monitoring by brain MRI at PML diagnosis
JC virus genotyping | 1 month, 3 months and 6 months
  JC virus genotyping in blood, cerebrospinal fluid (CSF) and urine by ultra-sensitive PCR at PML diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MARTIN-BLONDEL, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - CHU Bordeaux, Bordeaux
  - CHU Montpellier, Montpellier
  - CHU de TOULOUSE, Toulouse

IPD SHARING:
Plan to Share IPD: No